CLINICAL TRIAL: NCT00102544
Title: Electromagnetic Tracking of Devices During Interventional Procedures
Brief Title: Use of Tracking Devices to Locate Abnormalities During Invasive Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 050091; 05-CC-0091; NCT00671840 (obsolete NCT alias)
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-16

CONDITIONS: Adenocarcinoma; Prostate Neoplasms; Prostate Cancer; Renal Cell Carcinoma; Von Hippel Lindau Disease
Keywords: CT-Guided; Electromagnetic Tracking; Ultrasound-Guided Biopsy; Ablation; Surgical Navigation
MeSH Terms: conditions — Adenocarcinoma; Prostatic Neoplasms; Carcinoma, Renal Cell; von Hippel-Lindau Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All cohorts (prostate biopsy percutaneous biopsy and ablation) (Experimental): This study will consist of comparison of tracked imaging with near-simultaneous actual imaging .
  Interventions: Device: EM Tracking

INTERVENTIONS:
Device: EM Tracking — Utilizing electromagnetic tracking technology as a fusion and navigation tool for minimally invasive interventional procedures.

SUMMARY:
This study will evaluate the accuracy and effectiveness of an experimental tracking device for locating abnormalities during invasive procedures, such as biopsy or ablation, that cannot easily be visualized by usual imaging techniques, such as computed tomography (CT) scans or ultrasound. Some lesions, such as certain liver or kidney tumors, small endocrine abnormalities, and others, may be hard to find or only visible for a few seconds. The new method uses a needle with a miniature tracking device buried inside the metal that tells where the tip of the needle is located, somewhat like a mini GPS, or global positioning system. It uses a very weak magnet to localize the device like a miniature satellite system. This study will explore whether this system can be used in the future to more accurately place the needle in or near the desired location or abnormality.

Patients 18 years of age and older who have a lesion that needs to be biopsied or an ablation procedure that requires CT guidance may be eligible for this study. Candidates are screened with a medical history and review of medical records, including imaging studies.

Participants undergo the biopsy or ablation procedure as they normally would, with the following exceptions: some stickers are placed on the skin before the procedure and a very weak magnet is placed nearby. The needles used are similar to the ones that would normally be used except that they contain a metal coil or spring buried deep within the needle metal. The procedure involves the following steps:

1. Small 1-cm plastic donuts are place on the skin with tape.
2. A planning CT scan is done.
3. The CT scan is sent to the computer and matched to the patient's body location with the help of a very weak magnet.
4. The needle used for the procedure is placed towards the target tissue or abnormality and the "smart needle" location lights up on the old CT scan.
5. A repeat CT is done as it normally is to look for the location of the needle.
6. After the procedure the CT scans are examined to determine how well the new tool located the needle in the old scan.

DETAILED DESCRIPTION:
Background:

The effectiveness of targeting lesions or a specific area for surgery, angiography, CT-guided, or ultrasound-guided biopsy, or ablation, currently may be limited by the visibility of a target during the procedure. Accurate therapeutic intervention may depend upon accurate device placement, which may be very difficult in certain settings, such as when a liver tumor only is visible for a brief moment in time during the transient arterial phase of a contrast injection, soon disappearing on dynamic imaging. Surgery, angiography, image guided therapies and diagnostic procedures could be vastly improved by enabling the use of pre-procedural imaging during the procedure [such as location of difficult to visualize or transiently visible targets].Tracking devices allow the use of preoperative imaging during the procedure. Having this information available could vastly improve targeting accuracy of surgery, angiography, CT-guided, or ultrasound-guided biopsy or ablation.

A method of improving targeting could potentially benefit patients in the future by reducing total radiation exposure during CT scan or fluoroscopic monitoring of a biopsy, or decreasing certain surgical risks, although these are not specific subjects of this study. Various methods of device tracking have been used in the past throughout the 20th and 21st century in neurosurgery with the use of stereotactic frames for a similar purpose, to register pre-operative imaging to the patient during invasive procedures to guide treatment.

Objectives:

To define the clinical utility of electromagnetic tracking during interventional procedures in specific patient populations.

Eligibility:

1. All patients must have a CT, MR, or PET scan available in digital format.
2. Age greater than 18 years.
3. Patients must be actively enrolled on an NIH protocol and be scheduled for surgery, angiography, or CT- or ultrasound-guided biopsy.

Design:

This is an exploratory interventional study examining the use of a guidance system for navigating and monitoring devices like biopsy and ablation needles, ultrasound transducers, needle guides, guidewires, scalpels, and cauterization devices (herein referred to as device(s) ) for localization in relation to pre-operative images. There are 9 cohorts included in this protocol: The Open / Laparoscopic surgery and Angiography surgery cohorts are no longer open for accrual.

1. Prostate biopsy
2. Percutaneous biopsy for diagnostic correlation
3. percutaneous ablation for needle placement compilations
4. Open/Laparoscopic surgery
5. Angiography
6. Auto registration for biopsy
7. Auto registration for ablation
8. PET registration
9. prostate biopsy on which to determine the predictive value and relative strength of each MRI sequence in predicting cancer at a specific prostate core location.

The total accrual ceiling for this protocol is 3894 subjects.

All cohorts open for accrual are using exploratory interventions to define the specific patient population where fusion used during interventional procedures may have clinical value, and to characterize that clinical value in a specific patient population, such as but not limited to patients with specific regions of the prostate targeted, specific prostate volumes, prior negative prostate biopsies, or PSA values within a specific range.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission. Patient enrollment is by referral only.

1. All patients must have a pre-operative imaging (CT, MR, or PET scan) available in digital format.
2. Age greater than or equal to 18 years.
3. No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
4. The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.
5. All patients in non-prostate biopsy cohorts, must be undergoing an image-guided surgical or interventional radiology procedure such as an angiography or a CT/ US-guided biopsy as clinically indicated or IRB-approved under a separate research protocol.

PROSTATE BIOPSY COHORT (Cohorts 1 and 9) INCLUSION CRITERIA:

1. Patients are eligible if they have undergone a prostate MRI and have had abnormalities identified as follows:

1. PSA >2.5 OR abnormal digital rectal exam OR an abnormality identified on prostate MRI with a clinical indication for fusion biopsy
2. Pre-biopsy prostate MRI showing targetable lesions

EXCLUSION CRITERIA:

Patients with any of the following will be excluded from study entry:

1. Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study.
2. Patients unlikely able to hold reasonably still on a procedure table for the length of the procedure.
3. Inability to hold breath, if procedure will be performed with conscious sedation, and without general anesthesia.
4. Patients with pacemakers and other potentially electrically conductive implants.
5. Gross body weight above the CT table limit (606 pounds), if CT table used.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3894 (Estimated)
Dates: Start 2005-02-23 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using electromagnetic devices in different cohorts. | Day 1
  "TRE" Target Registration Error (distance between "virtual" needle position (tracking data) and the actual needle position ("CT" Computed Tomography confirmation scan))

SECONDARY OUTCOMES:
Success of ablation as determined by imaging | 3 months
  Primary effectiveness (success of ablation in local tumor control or success of biopsy in diagnostic biopsy sample). Successful ablation equals complete tumor ablation with a 5mm-1cm margin of normal tissue (if possible; quantified by the lack of enhancement of intravenous contrast material at 3 month follow up CT)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Seiler PG, Blattmann H, Kirsch S, Muench RK, Schilling C. A novel tracking technique for the continuous precise measurement of tumour positions in conformal radiotherapy. Phys Med Biol. 2000 Sep;45(9):N103-10. doi: 10.1088/0031-9155/45/9/402. PMID 11008969
- [Background] Frantz DD, Wiles AD, Leis SE, Kirsch SR. Accuracy assessment protocols for electromagnetic tracking systems. Phys Med Biol. 2003 Jul 21;48(14):2241-51. doi: 10.1088/0031-9155/48/14/314. PMID 12894982
- [Background] Solomon SB, White P Jr, Wiener CM, Orens JB, Wang KP. Three-dimensional CT-guided bronchoscopy with a real-time electromagnetic position sensor: a comparison of two image registration methods. Chest. 2000 Dec;118(6):1783-7. doi: 10.1378/chest.118.6.1783. PMID 11115473
- [Derived] Borde T, Varble NA, Hazen LA, Saccenti L, Garcia C, Digennaro M, Gurram S, Pinto PA, Turkbey B, Wood BJ. Impact of Discordance Between Magnetic Resonance Imaging and Ultrasound Volume Measurements on Prostate Fusion Biopsy Outcomes. J Urol. 2025 Apr;213(4):428-436. doi: 10.1097/JU.0000000000004368. Epub 2024 Dec 10. PMID 39657598
- [Derived] Ahdoot M, Lebastchi AH, Long L, Wilbur AR, Gomella PT, Mehralivand S, Daneshvar MA, Yerram NK, O'Connor LP, Wang AZ, Gurram S, Bloom J, Siddiqui MM, Linehan WM, Merino M, Choyke PL, Pinsky P, Parnes H, Shih JH, Turkbey B, Wood BJ, Pinto PA; Trio Study Group. Using Prostate Imaging-Reporting and Data System (PI-RADS) Scores to Select an Optimal Prostate Biopsy Method: A Secondary Analysis of the Trio Study. Eur Urol Oncol. 2022 Apr;5(2):176-186. doi: 10.1016/j.euo.2021.03.004. Epub 2021 Apr 10. PMID 33846112
- [Derived] Ahdoot M, Wilbur AR, Reese SE, Lebastchi AH, Mehralivand S, Gomella PT, Bloom J, Gurram S, Siddiqui M, Pinsky P, Parnes H, Linehan WM, Merino M, Choyke PL, Shih JH, Turkbey B, Wood BJ, Pinto PA. MRI-Targeted, Systematic, and Combined Biopsy for Prostate Cancer Diagnosis. N Engl J Med. 2020 Mar 5;382(10):917-928. doi: 10.1056/NEJMoa1910038. PMID 32130814
- [Derived] Siddiqui MM, Rais-Bahrami S, Turkbey B, George AK, Rothwax J, Shakir N, Okoro C, Raskolnikov D, Parnes HL, Linehan WM, Merino MJ, Simon RM, Choyke PL, Wood BJ, Pinto PA. Comparison of MR/ultrasound fusion-guided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. JAMA. 2015 Jan 27;313(4):390-7. doi: 10.1001/jama.2014.17942. PMID 25626035
- [Derived] Siddiqui MM, Rais-Bahrami S, Truong H, Stamatakis L, Vourganti S, Nix J, Hoang AN, Walton-Diaz A, Shuch B, Weintraub M, Kruecker J, Amalou H, Turkbey B, Merino MJ, Choyke PL, Wood BJ, Pinto PA. Magnetic resonance imaging/ultrasound-fusion biopsy significantly upgrades prostate cancer versus systematic 12-core transrectal ultrasound biopsy. Eur Urol. 2013 Nov;64(5):713-719. doi: 10.1016/j.eururo.2013.05.059. Epub 2013 Jun 12. PMID 23787357
- [Derived] Krucker J, Xu S, Venkatesan A, Locklin JK, Amalou H, Glossop N, Wood BJ. Clinical utility of real-time fusion guidance for biopsy and ablation. J Vasc Interv Radiol. 2011 Apr;22(4):515-24. doi: 10.1016/j.jvir.2010.10.033. Epub 2011 Feb 26. PMID 21354816
- [Derived] Krucker J, Xu S, Glossop N, Viswanathan A, Borgert J, Schulz H, Wood BJ. Electromagnetic tracking for thermal ablation and biopsy guidance: clinical evaluation of spatial accuracy. J Vasc Interv Radiol. 2007 Sep;18(9):1141-50. doi: 10.1016/j.jvir.2007.06.014. PMID 17804777
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-CC-0091.html